CLINICAL TRIAL: NCT06993727
Title: Prospective Study of Autoimmune Endocrine Disease-related Antibodies Before the Start of Immune Checkpoint Inhibitor Therapy
Brief Title: Autoimmune Endocrine Disease Related Antibodies Before the Start of Immune Checkpoint Inhibitor Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laura ICONARU (Other)
Responsible Party: Sponsor-Investigator, Laura ICONARU, Head of endocrinology clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUB-AC after ICI
Record Dates: First submitted 2025-05-19; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Autoimmunity
MeSH Terms: conditions — Autoimmune Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- immune checkpoint therapy (Experimental): The study aims to include all subjects eligible for immune checkpoint therapy at the participating study sites.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — For the analysis of the autoimmune endocrine disease related antibodies (Ab) before the start of the immunotherapy, a blood sample will be collected aligned with the first visit with the treating gastro-enterologist/oncologist/pneumologist for analysis of: anti-thyroglobulin Ab (aTg), anti-thyroperoxidase Ab (aTPO), TSH receptor antibodies (TRAb), pituitary Ab, adrenal Ab, and anti-glutamic acid decarboxylase (GAD) Ab.

SUMMARY:
Promising treatments have been added to the oncologist's arsenal in recent years. Treatments that, unlike conventional chemotherapy, do not aim to destroy cancer cells directly, but rather activate the patient's own immune system to recognize and attack tumor cells again. This new treatment is called immune checkpoint therapy. This involves administering antibodies (large Y-shaped proteins that can stick to the surface of cells) that remove the brakes from the immune system.

The disadvantage of this innovative treatment is that the rejuvenated immune system can also attack cells that we want it not to recognize - our own body's cells. This is called autoimmunity. Patients who receive immune checkpoint therapy may suffer from symptoms such as skin rashes, diarrhea, hepatitis or hypothyroidism.

The purpose of this study is to find biomarkers predictive of the development of these side effects, and possibly also predict a better outcome of the cancer therapy. The investigators will also look for the presence of antibodies against the endocrine glands (glands that produce hormones, such as the thyroid, adrenal, pituitary, and pancreas) before the start of the immune therapy.

DETAILED DESCRIPTION:
Immune checkpoint inhibitor therapy (ICI) is the current standard of care for many malignancies, due to its unique mechanism of action. These therapies release the brakes of the immune system by targeting cytotoxic T-lymphocyte antigen-4 (CTLA-4, e.g., ipilimumab, tremelimumab), programmed cell death-1 (PD-1, e.g., cemiplimab, dostarlimab, pembrolizumab, nivolumab) or its ligand (PD-L1, e.g., atezolizumab, avelumab, durvalumab). The flip side of the coin are immune-related adverse events (IrAE), including skin, intestinal and endocrinological toxicity, although any organ system can potentially be affected.

The prospective follow-up of the endocrine autoantibodies is an area of interest as the presence of thyroid autoantibodies is associated with the occurrence of thyroiditis with immunotherapy.

In turn, the occurrence of thyroiditis with immunotherapy is related to improved oncologic prognosis. Therefore, it would be of value to analyze whether the presence of thyroid autoimmunity (with positive thyroperoxidase and/or thyroglobulin autoantibodies) before the start of immunotherapy could be a marker of improved oncologic prognosis and outcome.

Furthermore, there is a gap in our knowledge of the impact of autoantibodies against less common endocrinopathies, such as hypophysitis (inflammation of the pituitary gland), adrenalitis (inflammation of the adrenal glands) or pancreas (type-1 like diabetes mellitus). Finding a prognostic factor for these types of endocrinopathy is equally important, as these patients may present with life-threatening endocrinopathy (adrenal crisis, diabetic ketoacidosis) and should be recognized and treated in a timely manner.

The main purpose of the current study is to evaluate the association between the autoimmune endocrine disease-related antibodies, the development of endocrine irAE and the impact on the tumor response including progression-free survival and overall survival.

For this study, the investigators aim to perform a blood sample before and during the immunotherapy, for the analysis of the autoimmune endocrine disease related antibodies (Ab): anti-thyroglobulin Ab (aTg), anti-thyroperoxidase Ab (aTPO), anti-TSH-receptor Ab (TSI), pituitary Ab, adrenal Ab, and anti-GAD. The included patients will be prospectively followed up.

ELIGIBILITY:
Inclusion Criteria:

* All subjects eligible for immune checkpoint therapy at the participating study sites. The cohort will consist of all subjects who consent to participate, and to use their information for future research and publication in a scientific journal.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Blood level of anti-thyroglobulin antibodies (aTg) | Baseline (before the start of the immunotherapy)
  Blood level of anti-thyroglobulin antibodies (aTg)
Blood level of anti-thyroglobulin antibodies (aTg) | 3 months after baseline
  Blood level of anti-thyroglobulin antibodies (aTg)
Blood level of anti-thyroglobulin antibodies (aTg) | 6 months after baseline
  Blood level of anti-thyroglobulin antibodies (aTg)
Blood level of anti-thyroperoxidase antibodies (aTPO) | Baseline (before the start of immunotherapy)
  Blood level of anti-thyroperoxidase antibodies (aTPO)
Blood level of anti-thyroperoxidase antibodies (aTPO) | 3 months after baseline
  Blood level of anti-thyroperoxidase antibodies (aTPO)
Blood level of anti-thyroperoxidase antibodies (aTPO) | 6 months after baseline
  Blood level of anti-thyroperoxidase antibodies (aTPO)
Blood levels of TSH receptor antibodies (TRAb) | Baseline (before the start of immunotherapy)
  Blood levels of TSH receptor antibodies (TRAb)
Blood levels of TSH receptor antibodies (TRAb) | 3 months after baseline
  Blood levels of TSH receptor antibodies (TRAb)
Blood levels of TSH receptor antibodies (TRAb) | 6 months after baseline
  Blood levels of TSH receptor antibodies (TRAb)
Blood level of pituitary antibody | Baseline (before the start of immunotherapy)
  Blood level of pituitary antibody
Blood level of pituitary antibody | 3 months after baseline
  Blood level of pituitary antibody
Blood level of pituitary antibody | 6 months after baseline
  Blood level of pituitary antibody
Blood level of adrenal antibody | Baseline (before the start of immunotherapy)
  Blood level of adrenal antibody
Blood level of adrenal antibody | 3 months after baseline
  Blood level of adrenal antibody
Blood level of adrenal antibody | 6 months after baseline
  Blood level of adrenal antibody
Blood level of anti-glutamic acid decarboxylase (GAD) antibody | Baseline (before the start of immunotherapy)
  Blood level of anti-glutamic acid decarboxylase (GAD) antibody
Blood level of anti-glutamic acid decarboxylase (GAD) antibody | 3 months after baseline
  Blood level of anti-glutamic acid decarboxylase (GAD) antibody
Blood level of anti-glutamic acid decarboxylase (GAD) antibody | 6 months after baseline
  Blood level of anti-glutamic acid decarboxylase (GAD) antibody

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen de Filette, MD, Study Director — CHU Brugmann
Locations (3):
- Belgium (3):
  - C.H.U. Saint-Pierre, Brussels
  - CHU Brugmann, Brussels
  - HUB - Institut Jules Bordet, Brussels

IPD SHARING:
Plan to Share IPD: No